CLINICAL TRIAL: NCT03795571
Title: Lenalidomide, Rituximab, Gemcitabine, Oxaliplatin and Dexamethasone (R2-GOD) in Treatment of Relapse/Refractory DLBCL:A Phase I Study
Brief Title: Lenalidomide, Rituximab, Gemcitabine, Oxaliplatin and Dexamethasone in Relapse and Refractory DLBCL
Acronym: R2-GOD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2-GOD regimen
Record Dates: First submitted 2019-01-01; First posted 2019-01-07 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Diffuse Large B-cell Lymphoma Recurrent; Diffuse Large B Cell Lymphoma Refractory
Keywords: lenalidomide; R-GOD; DLBCL
MeSH Terms: interventions — Rituximab; Gemcitabine; Oxaliplatin; Dexamethasone; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R2-GOD (Experimental)
  Interventions: Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Dexamethasone; Drug: Lenalidomide Oral Capsule

INTERVENTIONS:
Drug: Rituximab — Rituximab 375mg/m2，d0
Drug: Gemcitabine — Gemcitabine 1000mg/m2，d1，d5
Drug: Oxaliplatin — Oxaliplatin 75mg/m2，d1
Drug: Dexamethasone — Dexamethasone 40mg/d，d1~d4
Drug: Lenalidomide Oral Capsule — Lenalidomide 10mg/d、15mg/d、20mg/d、25mg/d d1~d10； 21days a cycle

SUMMARY:
Previous study showed that Lenalidomide or R-GDP could achieve response in Relapse and Refractory DLBCL.The investigators therefore design this phase I study to investigate the safety and efficacy of R2-GOD in relapsed diffuse large-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old;
* ECOG PS 0- 2;
* Histologically confirmed diffuse large B cell lymphoma（With exception of Primary mediastinal large B cell lymphoma、Primary central nervous system lymphoma、HIV-related lymphoma),relapse or refractory,defined as:

  * relapse after standard first-line immunochemotherapy( R-CHOP or R-CHOP like)
  * SD as best response after 4 cycles or PD after 2 cycles of first-line immunochemotherapy;
* a measurable or evaluable disease at the time of enrollment(diameter ≥ 1.5cm）；
* Eligible for subsequent autologous stem cell transplantation；
* Female subjects in childbearing age, their serum or urine pregnancy test must be negative. All patients must agree to take effective contraceptive measures during the trial measures
* Expected survival ≥ 12 weeks；
* Understand and voluntarily sign an informed consent form, able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Women who are pregnant or lactating. Patients have breeding intent in 12 months or cannot take effective contraceptive measures during the trial measures；
* Uncontrollable active infection within four week. Prophylactic antibiotic, antiviral and antifungal treatment is permissible. Active hepatitis B or hepatitis C virus infection, as well as acquired, congenital immune deficiency diseases, including but not limited to HIV-infected persons；
* Used of systemic anti-tumor treatment within four weeks；
* CNS or meningeal involvement;
* Poor hepatic and/or renal function, defined as total bilirubin, ALT, AST, Cr more than two fold of upper normal level,Ccr< 50 mL/min unless these abnormalities were related to the lymphoma;
* Poor bone-marrow reserve, defined as neutrophil count less than 1.5×10⁹/L or platelet count less than 75×10⁹/L, unless caused by bone marrow infiltration;
* New York Heart Association class III or IV cardiac failure; or Ejection fraction less than 50%;or history of following disease in past 6 months: acute coronary syndrome、acute heart failure、severe ventricular arrhythmia；
* Known sensitivity or allergy to investigational Product;
* Major surgery within three weeks;
* Presence of Grade III nervous toxicity within past two weeks;
* Active and severe infectious diseases;
* History of DVT or PE within past 12 months；
* Any potential drug abuse, medical, psychological or social conditions which may disturb this investigation and assessment;
* In any conditions which investigator considered ineligible for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose and dose limited toxicity | 28 days after first cycle of R2-GOD regimen

SECONDARY OUTCOMES:
Overall response rate, | 6 months
  overall response rate after treated by R-GemOx or R-miniCHOP overall response rate after treated by R2-GOD regimen regimen
Progressive free survival | 2 years
  from date of inclusion to date of progression, relapse, or death from any causePFS：from date of inclusion to date of progression, relapse, or death from any cause
Overall survival | 2 years
  from the date of inclusion to date of death, irrespective of cause

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, PhD& MD, Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital)
Locations (1):
- The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feldman T, Mato AR, Chow KF, Protomastro EA, Yannotti KM, Bhattacharyya P, Yang X, Donato ML, Rowley SD, Carini C, Valentinetti M, Smith J, Gadaleta G, Bejot C, Stives S, Timberg M, Kdiry S, Pecora AL, Beaven AW, Goy A. Addition of lenalidomide to rituximab, ifosfamide, carboplatin, etoposide (RICER) in first-relapse/primary refractory diffuse large B-cell lymphoma. Br J Haematol. 2014 Jul;166(1):77-83. doi: 10.1111/bjh.12846. Epub 2014 Mar 25. PMID 24661044
- [Background] Martin A, Redondo AM, Dlouhy I, Salar A, Gonzalez-Barca E, Canales M, Montes-Moreno S, Ocio EM, Lopez-Guillermo A, Caballero D; Spanish Group for Lymphomas and Autologous Bone Marrow (GELTAMO). Lenalidomide in combination with R-ESHAP in patients with relapsed or refractory diffuse large B-cell lymphoma: a phase 1b study from GELTAMO group. Br J Haematol. 2016 Apr;173(2):245-52. doi: 10.1111/bjh.13945. Epub 2016 Feb 5. PMID 26847165
- [Background] Crump M, Kuruvilla J, Couban S, MacDonald DA, Kukreti V, Kouroukis CT, Rubinger M, Buckstein R, Imrie KR, Federico M, Di Renzo N, Howson-Jan K, Baetz T, Kaizer L, Voralia M, Olney HJ, Turner AR, Sussman J, Hay AE, Djurfeldt MS, Meyer RM, Chen BE, Shepherd LE. Randomized comparison of gemcitabine, dexamethasone, and cisplatin versus dexamethasone, cytarabine, and cisplatin chemotherapy before autologous stem-cell transplantation for relapsed and refractory aggressive lymphomas: NCIC-CTG LY.12. J Clin Oncol. 2014 Nov 1;32(31):3490-6. doi: 10.1200/JCO.2013.53.9593. Epub 2014 Sep 29. PMID 25267740
- [Background] Shen QD, Zhu HY, Wang L, Fan L, Liang JH, Cao L, Wu W, Xia Y, Li JY, Xu W. Gemcitabine-oxaliplatin plus rituximab (R-GemOx) as first-line treatment in elderly patients with diffuse large B-cell lymphoma: a single-arm, open-label, phase 2 trial. Lancet Haematol. 2018 Jun;5(6):e261-e269. doi: 10.1016/S2352-3026(18)30054-1. Epub 2018 May 8. PMID 29752199